CLINICAL TRIAL: NCT02799953
Title: Evaluating a Technology-augmented Self-monitoring Model for Glycemic and Blood Pressure Control and Medication Adherence in Type 2 Diabetes and Hypertension Patients: a Randomized Controlled Trial
Brief Title: Technology-augmented Self-monitoring Model Among Patients With Type 2 Diabetes and Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Calvin Or, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HMRF12133231
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
Keywords: diabetes mellitus and hypertension; consumer health information technology; self-monitoring; randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Technology-based self-management model (Experimental): Participants randomized to the intervention group will be given a tablet-based, interactive touch-screen self-monitoring system free of charge to perform disease self-monitoring in their homes.
  Interventions: Device: Technology-based self-management model
- Conventional self-management (No Intervention): Participants randomized to the usual care group will not be provided access to tablet computers but a 2-in-1 blood pressure and blood glucose monitor and a paper-based log book to perform conventional self-monitoring.

INTERVENTIONS:
Device: Technology-based self-management model — Participants in the technology-augmented self-monitoring model (intervention group) will use a tablet-based, interactive touch screen self-monitoring system to monitor and manage their chronic conditions. The system is designed to augment patients' abilities to assess, record, and review their health signs while providing text-, audio-, and video-based resources supporting disease self-care.
  Arms: Technology-based self-management model

SUMMARY:
Objective: To develop and evaluate a technology-augmented self-monitoring model using a randomized controlled trial to demonstrate whether patients with co-morbid type 2 diabetes mellitus and hypertension can improve their glycemic and blood pressure control, adherence to medication regimens, and other relevant outcomes by using a tablet-based consumer health information technology (CHIT) to support the self-monitoring and self-management of their chronic conditions.

Design: A two-group, randomized controlled trial with follow-up assessments 8, 12, 16, and 24 weeks after the baseline evaluation.

Setting: Patients' homes.

Participants: Two hundred and ninety-six adult patients with type 2 diabetes mellitus and hypertension who receive their health care from a local community health service network or a major hospital will be recruited.

Interventions: Participants in the technology-augmented self-monitoring model (intervention group) will use a tablet-based, interactive touch screen self-monitoring system to monitor and manage their chronic conditions. The system is designed to augment patients' abilities to assess, record, and review their health signs while providing text-, audio-, and video-based resources supporting disease self-care. The participants in the usual-care group will perform conventional self-monitoring.

Outcome measures: The primary outcomes will be glycemic control measured by changes in HbA1c,blood pressure control assessed by changes in systolic and diastolic blood pressure, and medication compliance. The secondary outcomes will be adherence to diabetes and hypertension self-care activities and knowledge of diabetes and hypertension.

Implication: This study will improve our understanding of the clinical value of CHITs in chronic disease self-monitoring and self-management.

DETAILED DESCRIPTION:
Subject recruitment: The person-in-charge/managers of the departments of the hospitals/the health service centers will go through the in-house medical documents to identify adults with a diagnosis of type 2 diabetes and hypertension and invite them to attend an information session, in which the project's lead PI (Dr. Calvin Or) and research assistants will introduce the study; determine their eligibility based on their self-reported demographic data, health information, and/or medical records; and collect their contact information. Later, the research assistant will telephone the eligible patients to schedule a first visit to their homes for enrollment.

Intervention: The participants randomized to the intervention group will be given a tablet-based, interactive touch-screen self-monitoring system free of charge to perform disease self-monitoring in their homes. The objectives of the system are to empower patients' ability to self-monitor and improve their self-care adherence and medication compliance by enabling access to various e-support, information, resources, and self-monitoring tools in a timely manner. It runs on a 10-inch touch-screen tablet computer that is programmed to connect to a 2-in-1 blood pressure and glucose monitor. Measurement modules are available for assessing and recording blood pressure, pulse, and blood glucose level. The assessment records are fully automated and can be retrieved and reviewed in structured tables and charts. Patients can determine whether assessment values that deviate from the critical levels may need attention based on the "normal value ranges" indicated by the system. The system also has a module that provides both text- and video-based learning resources related to the causes and prevention of type 2 diabetes and hypertension, self-care, salt and sodium intake, diet, action plan (e.g., appropriate actions in response to symptoms), exercise, and stress management. The care information and video capability allow patients to easily learn how to self-monitor and self-manage. In addition, the system has a reminder function that can be programmed to emit audible reminders at predetermined times alerting patients to take their prescribed medications. A secured web portal (http://selfcare.imse.hku.hk/) is available for authorized, non-patient users such as caregivers and families to remotely review and monitor the assessment values of key patient health signs using their own mobile devices or computers.

Randomization: Participants will be stratified into four groups based on the HbA1c and systolic blood pressure measurements: (i) HbA1c ≤ 8% and systolic BP ≤ 159 mm Hg, (ii) HbA1c ≤ 8% and systolic BP ≥ 160 mm Hg, (iii) HbA1c > 8% and systolic BP ≤ 159 mm Hg, and (iv) HbA1c > 8% and systolic BP ≥ 160 mm Hg. These cut-offs for grouping were set based on previous studies (2, 3) and clinical judgement. Within each stratum, the patients will be block-randomized into the study groups using randomly permuted blocks and sequentially numbered, opaque, sealed envelopes. The randomization and allocation process will be based on the practical guide for permuted blocks randomization in a stratified trial, as described in Doig and Simpson (4), and handled centrally by a researcher in response to a telephone call.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* with a physician-confirmed diagnosis of type 2 diabetes and hypertension of at least 1 month's duration
* normal (or corrected-to-normal) vision
* no cognitive or physical impairment
* ability to perform disease self-monitoring and self-management
* a willingness to use the tablet self-monitoring system
* the ability to understand written and spoken Chinese

Exclusion Criteria:

* with abnormal vision and physical impairments
* with any unstable or life-threatening illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
changes in HbA1c | from baseline to 12 and 24 weeks
changes in systolic and diastolic blood pressure | from baseline to 8, 16, and 24 weeks

SECONDARY OUTCOMES:
medication adherence | from baseline to 8, 16, and 24 weeks
adherence to diabetes self-care activities | from baseline to 8, 16, and 24 weeks
adherence to hypertension self-care activities | from baseline to 8, 16, and 24 weeks
changes in answering diabetes knowledge questions | from baseline to 8, 16, and 24 weeks
changes in answering hypertension knowledge questions | from baseline to 8, 16, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Or, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Pamela Youde Nethersole Eastern Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Or C, Tao D. Usability study of a computer-based self-management system for older adults with chronic diseases. JMIR Res Protoc. 2012 Nov 8;1(2):e13. doi: 10.2196/resprot.2184. PMID 23612015
- [Background] Green BB, Cook AJ, Ralston JD, Fishman PA, Catz SL, Carlson J, Carrell D, Tyll L, Larson EB, Thompson RS. Effectiveness of home blood pressure monitoring, Web communication, and pharmacist care on hypertension control: a randomized controlled trial. JAMA. 2008 Jun 25;299(24):2857-67. doi: 10.1001/jama.299.24.2857. PMID 18577730
- [Background] McMahon GT, Gomes HE, Hickson Hohne S, Hu TM, Levine BA, Conlin PR. Web-based care management in patients with poorly controlled diabetes. Diabetes Care. 2005 Jul;28(7):1624-9. doi: 10.2337/diacare.28.7.1624. PMID 15983311
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Derived] Or CK, Liu K, So MKP, Cheung B, Yam LYC, Tiwari A, Lau YFE, Lau T, Hui PSG, Cheng HC, Tan J, Cheung MT. Improving Self-Care in Patients With Coexisting Type 2 Diabetes and Hypertension by Technological Surrogate Nursing: Randomized Controlled Trial. J Med Internet Res. 2020 Mar 27;22(3):e16769. doi: 10.2196/16769. PMID 32217498